CLINICAL TRIAL: NCT04131127
Title: Cerebral Protection of Acute Embolic Burden During Transcatheter Aortic Valve Implantation in Low Risk Patients
Brief Title: Sentinel Low Risk Registry
Status: Completed | Type: Observational
Sponsor: CVPath Institute Inc. (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CP2561-0316
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — We will collect debris that have been captured in the Sentinel filter and perform pathology on those specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Sentinel Device — Sentinel Device used during TAVI in a Low Risk Patient

SUMMARY:
This registry is designed to quantify embolic debris capture rate in patients at low surgical risk treated with the Sentinel System during TAVI.

DETAILED DESCRIPTION:
The SENTINEL-LIR Study is a multicenter, prospective registry to observe rate and type of debris capture in subjects at low surgical risk undergoing TAVI to demonstrate the positive effects of the use of the Sentinel System. Histopathology of captured debris from the Sentinel System will be analyzed.

The primary objective is to determine the presence or absence of particles of 7 discreet tissue types: acute thrombus (with or without associated tissue/foreign material), organizing thrombus, valve tissue, arterial wall/necrotic core, calcification, foreign material, and myocardium. Morphometric assessment of the debris (sizes >150 m, >500 m, and >1,000 m).

Patients will be screened for inclusion and exclusion criteria and documents which will have been reviewed and approved by the local Ethics Committee or regulatory authority prior to undergoing any study related exams or procedures.

Fifty (50) subjects will be enrolled in the study from an estimated 6 different sites.

ELIGIBILITY:
Inclusion Criteria:

1. Severe symptomatic aortic valve stenosis
2. Planned use of Sentinel System
3. Subject planned for transfemoral TAVI with valve system approved by U.S. FDA for low risk patients
4. STS-PROM score of less than 4% and agreement by Heart Team that patients meet criteria for low surgical risk

Exclusion Criteria:

1. Current or recent cerebrovascular accident (stroke, TIA) <6 months
2. Transapical, direct aortic or subclavian TAVI access
3. Carotid stenting or endarterectomy in last 6 weeks
4. Prior aortic valve replacement
5. Concomitant procedure with TAVI such as CABG, PCI, etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is comprised of subjects with severe native aortic valve stenosis who meet the commercially approved indications for TAVI and comply with the inclusion/exclusion criteria described below.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
The SENTINEL-LIR Study | 12 months
  To determine the incidence and type of debris capture in SENTINEL devices deployed during TAVI in patients at low surgical risk

CONTACTS AND LOCATIONS:
Overall Officials: Aloke V Finn, MD, Principal Investigator — CVPath Institute
Locations (4):
- United States (4):
  - Columbia University Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Pinnacle, Wormleysburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Seeger J, Kapadia SR, Kodali S, Linke A, Wohrle J, Haussig S, Makkar R, Mehran R, Rottbauer W, Leon M. Rate of peri-procedural stroke observed with cerebral embolic protection during transcatheter aortic valve replacement: a patient-level propensity-matched analysis. Eur Heart J. 2019 May 1;40(17):1334-1340. doi: 10.1093/eurheartj/ehy847. PMID 30590554
- [Background] Schmidt T, Leon MB, Mehran R, Kuck KH, Alu MC, Braumann RE, Kodali S, Kapadia SR, Linke A, Makkar R, Naber C, Romero ME, Virmani R, Frerker C. Debris Heterogeneity Across Different Valve Types Captured by a Cerebral Protection System During Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2018 Jul 9;11(13):1262-1273. doi: 10.1016/j.jcin.2018.03.001. PMID 29976363
- [Background] Lazar RM, Pavol MA, Bormann T, Dwyer MG, Kraemer C, White R, Zivadinov R, Wertheimer JC, Thone-Otto A, Ravdin LD, Naugle R, Mechanic-Hamilton D, Garmoe WS, Stringer AY, Bender HA, Kapadia SR, Kodali S, Ghanem A, Linke A, Mehran R, Virmani R, Nazif T, Parhizgar A, Leon MB. Neurocognition and Cerebral Lesion Burden in High-Risk Patients Before Undergoing Transcatheter Aortic Valve Replacement: Insights From the SENTINEL Trial. JACC Cardiovasc Interv. 2018 Feb 26;11(4):384-392. doi: 10.1016/j.jcin.2017.10.041. Epub 2018 Feb 1. PMID 29397361
- [Background] Kapadia SR, Kodali S, Makkar R, Mehran R, Lazar RM, Zivadinov R, Dwyer MG, Jilaihawi H, Virmani R, Anwaruddin S, Thourani VH, Nazif T, Mangner N, Woitek F, Krishnaswamy A, Mick S, Chakravarty T, Nakamura M, McCabe JM, Satler L, Zajarias A, Szeto WY, Svensson L, Alu MC, White RM, Kraemer C, Parhizgar A, Leon MB, Linke A; SENTINEL Trial Investigators. Protection Against Cerebral Embolism During Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2017 Jan 31;69(4):367-377. doi: 10.1016/j.jacc.2016.10.023. Epub 2016 Nov 1. PMID 27815101
- [Derived] Kawakami R, Gada H, Rinaldi MJ, Nazif TM, Leon MB, Kapadia S, Krishnaswamy A, Sakamoto A, Sato Y, Mori M, Kawai K, Cornelissen A, Park JE, Ghosh SKB, Abebe BG, Romero M, Virmani R, Finn AV. Characterization of Cerebral Embolic Capture Using the SENTINEL Device During Transcatheter Aortic Valve Implantation in Low to Intermediate-Risk Patients: The SENTINEL-LIR Study. Circ Cardiovasc Interv. 2022 Apr;15(4):e011358. doi: 10.1161/CIRCINTERVENTIONS.121.011358. Epub 2022 Mar 11. No abstract available. PMID 35272475